CLINICAL TRIAL: NCT06009159
Title: Vagus Nerve Stimulation(VNS) As Treatment For Fibromyalgia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lucy Chen, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023P001211
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Fibromyalgia
Keywords: Vagus nerve stimulation,; pain; fibromyalgia symptoms
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Intervention Model Description: 4-week of clinical study with a total of 60 subjects, randomized into 2 groups (30 subjects in tVNS and 30 subjects in control group )
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcutaneous Vagus Nerve Stimulation(tVNS) (Experimental): receive tVNS 30 minutes per session, twice/day for 4 weeks and maintain regular medication treatment without change.
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation
- Sham Control group (No Intervention): receive sham point stimulation 30 minutes per session, twice/day for 4 weeks and maintain regular medication treatment without change.

INTERVENTIONS:
Device: Transcutaneous Vagus Nerve Stimulation — 30 minutes stimulation, twice per day for 4 weeks
  Arms: Transcutaneous Vagus Nerve Stimulation(tVNS)

SUMMARY:
Fibromyalgia (FM) is a syndrome with clinical symptoms involving multiple systems. The efficacy of current treatments is inadequate, and more alternative modalities are needed for the management of FM patients. The parasympathetic vagus nerve innervates and integrates sensory, motor, and autonomic systems and has been suggested to play a role in pain modulation. The role of vagus nerve stimulation (VNS) as a treatment option for FM patients is yet to be investigated. The investigators propose to examine the hypothesis that vagus nerve stimulation could improve pain and related comorbid symptoms for FM patients.

DETAILED DESCRIPTION:
The main goal of this study is to generate preliminary data on the effect of VNS on FM symptoms. Specifically, the investigators will utilize a recently developed, non-invasive method of tVNS (transcutaneous VNS) via auricular branches of vagus nerve (ABVN). The investigators plan to conduct an 4-week clinical study with 60 subjects randomized into 2 groups(tVNS group and control group; 30 subjects in each group). The primary outcome measure will be pain intensity. The secondary outcome measures will be fatigue, sleep, and other health-related quality of life measure. These outcome measures will be made at baseline week 0 (before any intervention), and at the end of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 to 80 years old, including both male and female subjects.
2. Subject has a documented diagnosis of FM for at least three months. This requirement is to avoid the uncertainty of an unstable pain condition and to minimize the study variation.
3. Subject has a pain score of 4 or above (numeric pain score: 0 - 10 from no pain to worst pain).

Exclusion Criteria:

1. Subject has current cardiac arrhythmia or had implanted cardiac pacemaker or AICD device.
2. Subject has major psychiatric disorder required hospitalization in the last 3 months.
3. Subject has active infection at the site of device application.
4. Subject has recurrent syncope symptoms within the past three months.
5. Subject is pregnant.
6. Subject has had VNS treatment within the past two months.

   .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
A modified McGill Pain Questionnaire | at 0,4, weeks of the study,
  Pain intensity, 0-10 score, with 0 means no pain and 10 means worst pain

SECONDARY OUTCOMES:
Multidimensional Fatigue Inventory | at 0,4,8 weeks of the study
  Fatigue level, 1-5 score, base on the statement, answer 1 means completely true and answer 5 means no, that is not true.
Medical Outcomes Study Sleep Scale | at 0,4,8 weeks of the study
  sleep quality, score 1-6, base on the statement, answer 1 means all of the time, answer 6 means none of the time
Revised Fibromyalgia Impact Questionnaire | at 0,4,8 weeks of the study
  Fibromyalgia impact, 0-10, answer 0 means no impact, 10 means the most impact
Medical Outcomes Study Questionnaire Short Form 36 | at 0, 4, 8 weeks of the study
  Quality of life measure, answer in descriptive degree of impact to life from: not at all, slightly, moderately, severe, very severe.
Blood inflammation marker | at 0, 4, 8 weeks of the study
  collect blood sample for cytokines level
Assessment of gut microbiome changes through genomic phenotypic | at 0, 4, 8 weeks of the study
  collect stool sample to analyze bacterial composition and metabolomic profiles of gut microbiome

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moisset X, Lanteri-Minet M, Fontaine D. Neurostimulation methods in the treatment of chronic pain. J Neural Transm (Vienna). 2020 Apr;127(4):673-686. doi: 10.1007/s00702-019-02092-y. Epub 2019 Oct 21. PMID 31637517
- [Background] Yuan H, Silberstein SD. Vagus Nerve and Vagus Nerve Stimulation, a Comprehensive Review: Part I. Headache. 2016 Jan;56(1):71-8. doi: 10.1111/head.12647. Epub 2015 Sep 14. PMID 26364692
- [Background] Maffei ME. Fibromyalgia: Recent Advances in Diagnosis, Classification, Pharmacotherapy and Alternative Remedies. Int J Mol Sci. 2020 Oct 23;21(21):7877. doi: 10.3390/ijms21217877. PMID 33114203